CLINICAL TRIAL: NCT02798328
Title: Direct Oral Anticoagulant Assay Detection & Classification Study for the TEG 6S System
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100394
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: DOAC Eligible Subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Reference Range: Healthy Subjects
  Interventions: Device: TEG6s DOAC Cartridge
- DOAC Pivotal: DOAC Eligible Subjects
  Interventions: Device: TEG6s DOAC Cartridge

INTERVENTIONS:
Device: TEG6s DOAC Cartridge — Testing subjects for presence of DOAC

SUMMARY:
Observational trial to evaluate the effectiveness of the TEG6s DOAC cartridge to detect and classify the presence of DOAC drugs in a subject.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* DOAC administered for a minimum of 7 days

Exclusion Criteria:

* Genetic Bleeding disorders. Known or subsequently discovered inherited defects of coagulation (e.g. hemophilia or Von Willebrand disease)
* Not known when last two DOAC doses were administered prior to blood draw
* DOAC first administered (or resumed after temporary cessation) less than 7 days prior to blood draw
* DOAC dosage outside of manufacturer's recommended range (e.g. study subject with renal impairment and supratherapeutic dose)
* Heparin or LMWH administered within 7 days prior to blood draw
* On any medications known to affect coagulation status and listed below
* Bruising, wounds or scarring in the area of venipuncture

List of medications known to affect coagulation status

1. Vitamin K Antagonists [VKAs] Warfarin Phenprocoumon Acenocoumarol Tecarfarin [ATI-5923] Phenindione Anisindione Elinogrel Vorapaxar Atopaxar
2. Heparin and Heparins Unfractionated Heparin [UFH] LMWH Fondaparinux Idraparinux Danaparoid
3. Vasopressin Analogues DDAVP
4. Direct Thrombin [IIa] Inhibitors Hirudin Lepirudin Bivalirudin Argatroban
5. Defibrinating Agents Ancrod

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DOAC Eligible Subjects
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Presence / Absence of DOAC Drug | 1 week

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Memorial Hospital South Bend, South Bend, Indiana
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Inova Health Care Services, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Undecided